CLINICAL TRIAL: NCT01526044
Title: Continuous Glucose Monitoring by Subcutaneous Measurement Compared to Frequent Point of Care Measurement by Accu Chek in Critically Ill Patients; a Randomized Controlled Trial (RESCUEII)
Brief Title: Continuous Glucose Monitoring by Subcutaneous Measurement Compared to Frequent Point of Care Measurement by Accu Chek in Critically Ill Patients
Acronym: RESCUEII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, PHJ van der Voort, PHJ van der Voort, MD, PhD, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL33495.100.10
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Hyperglycaemia; Hypoglycaemia
Keywords: hyperglycemia; hypoglycemia; insulin; critical illness; intensive insulin therapy; continuous glucose monitoring; CGM; interstitial fluid glucose; intensive care unit; Blood glucose
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia; Insulin Resistance; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Freestyle group (Experimental): Glucose levels are being monitored with the Freestyle Navigator up to 5 days, or until discharge from the ICU
  Interventions: Device: Freestyle Navigator
- AccuChek group (Active Comparator): Glucose levels are being measured by the AccuChek. Patients also get a Freestyle Navigator, which will be blinded. The device will stay on the patient up to 5 days, or until discharge from the ICU.
  Interventions: Device: Freestyle Navigator

INTERVENTIONS:
Device: Freestyle Navigator — Continuous glucose monitoring by subcutaneous measurement in the interstitial fluid
  Other Names: Freestyle Navigator, Abbott Diabetes Care

SUMMARY:
The purpose of this study is to evaluate the accuracy and reliability of the continuous glucose monitoring system the FreeStyle Navigator® (Abbott, Diabetes Care) in critically ill patients by comparing subcutaneous measuring with the current standard of arterial measuring by a point of care glucometer.

DETAILED DESCRIPTION:
Most patients admitted to the ICU are treated with intensive insulin therapy, according to a locally developed glucose treatment protocol. The use of a continuous glucose monitoring in critically ill patients could have the following advantages:

* Better insight in the alterations of the blood glucose levels
* Early detection of hypoglycemia's or hyperglycaemia's, and subsequently more stable glycemic levels.
* Fewer blood samples
* Decreased workload for the nursing staff

In this study, patients will be randomized in: 1. The Freestyle group or 2. The AccuChek Group.

Patients in both groups will receive a Freestyle Navigator device, which will stay on the patient up to 5 days, or until discharge from the ICU.

The medical treatment of both study groups will be equal, except for the frequency of the glucose level measurements and the resulting adjustments according to the treatment protocol. In the Freestyle group extra glucose level measurements will be made in response to alarms from the device.

In both groups, every 4 hours blood glucose values will be obtained using a blood gas analyzer (BGA). When a control measurement by BGA results in a glucose level of <2.2 or >25 mmol/l, the value will be transmitted to the Patient Data Management System (PDMS) and gives an alarm. Otherwise, the value will be blinded in the PDMS.

Freestyle Navigator data will be downloaded from the device. Blood glucose values obtained in the course of usual care will be compared with time-matched Freestyle Navigator values to assess device accuracy.

ELIGIBILITY:
Inclusion Criteria:

* ICU-patients > 18 years
* Expected length of stay on the ICU > 24 hours
* Indication for glucose regulation with insulin (according to the current glucose treatment protocol)
* Availability of the Freestyle Navigator

Exclusion Criteria:

* Participation in another trial subject to the WMO
* Lack of informed consent
* Contraindication for the use of the Accu Chek (for example peritoneal dialysis, Ht <0,20 of > 0,65; paracetamol intoxication)
* Contraindication for placement of the subcutaneous glucose sensor
* Participation in this trial during previous ICU admittance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of severe hyperglycaemias and hypoglycaemias with blood glucose levels >25 mmol/l and <2.2 mmol/l

SECONDARY OUTCOMES:
Time duration that the blood glucose levels of a patient are within the 'target range' (measured with the freestyle Navigator®)
  The target range in the ICU of the OLVG is set between 5 and 9 mmol/l according to the local treatment protocol
Time duration that the blood glucose levels of a patient are under and above the 'target range' (measured with the freestyle Navigator®)
  The target range in the ICU of the OLVG is set between 5 and 9 mmol/l according to the local treatment protocol
- Variability of the glycemic levels by arterial measuring with the blood gas analyzer (BGA), determined by the Mean Absolute Glucose change per hour (MAG)
  Mean Absolute Glucose change per hour:
  ΔBGA / Δtime The MAG is calculated by taking the sum of all absolute glucose changes during admission (measured by BGA) and dividing this by the total time spent in the ICU in hours.
Length of stay in the ICU
Mortality
False positive frequency of alarms of the Freestyle Navigator®
  Verified by the glucose level measurements by blood gas analyzer
Number of undesirable low glucose levels per 24 hours | 24 hours
  blood glucose levels between 2,5 and 5 mmol/l
Number of missed hypoglycemia's with the AccuChek (measured with the Freestyle Navigator®)
Number of blood samples per day | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: P HJ van der Voort, MD, PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands

REFERENCES:
- [Derived] Boom DT, Sechterberger MK, Rijkenberg S, Kreder S, Bosman RJ, Wester JP, van Stijn I, DeVries JH, van der Voort PH. Insulin treatment guided by subcutaneous continuous glucose monitoring compared to frequent point-of-care measurement in critically ill patients: a randomized controlled trial. Crit Care. 2014 Aug 20;18(4):453. doi: 10.1186/s13054-014-0453-9. PMID 25139609